CLINICAL TRIAL: NCT07100067
Title: A Clinical Study to Evaluate the Safety, Tolerance and Efficacy of LCAR- F33S Cell Therapy in Patients With Relapsed/Refractory Multiple Myeloma.
Brief Title: LCAR-F33S in Treatment of Relapsed/Refractory Multiple Myeloma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Legend Biotech Co. (Industry)
Collaborators: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB2502-0001
Record Dates: First submitted 2025-07-30; First posted 2025-08-03 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Relapsed/Refractory Multiple Myeloma(MM)
Keywords: multiple myeloma; Relapsed/Refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Single Group Assignment ，LCAR-F33S cells intravenous infusion Pretreatment of cyclophosphamide and fludarabine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LCAR-F33S (Experimental): Each subject will be given a single-dose LCAR- F33S cells infusion at each dose level.
  Interventions: Biological: LCAR- F33S cells intravenous infusion

INTERVENTIONS:
Biological: LCAR- F33S cells intravenous infusion — Prior to infusion of the LCAR- F33S cell, Subjects will receive a conditioning premedication regimen consisting of cyclophosphamide and fludarabine.

SUMMARY:
A prospective, single-arm, open-label dose-exploration and expansion study to evaluate the safety, tolerability, pharmacokinetics, and antitumor efficacy characteristics of LCAR-F33S in patients with relapsed/refractory multiple myeloma(Investigator-initiated Study).

DETAILED DESCRIPTION:
This study is a prospective, single-arm, open-label clinical study to evaluate the safety, tolerability, pharmacokinetics, and antitumor efficacy characteristics of LCAR-F33S in patients with relapsed/refractory multiple myeloma. All subjects who meet the eligibility criteria will receive intravenous injection of LCAR-F33S cell injection. The study will include the following sequential phases: screening, apheresis, pre-treatment (lymphodepleting chemotherapy), treatment, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in clinical research.
* Age ≥18 years old.
* Eastern Cooperative Oncology Group (ECOG) score 0-2.
* Examination evidence of initial diagnosis of MM according to IMWG diagnostic criteria.
* Measurable lesions were present.
* Subjects have received treatment with one PI, one IMiD and a CD38 monoclonal antibody.
* Subjects have received at least three previous lines of multiple myeloma therapy, each with at least one complete therapy cycle, unless the best response to the therapeutic regimen was documented as disease progression (PD confirmed according to IMWG criteria).
* Expected survival ≥3 months.
* Clinical laboratory values in the screening period meet criteria.

Exclusion Criteria:

* Received previous therapy targeting FcRH5 targets.
* Prior antineoplastic therapy and meet exclusion criteria (before apheresis);
* Subjects had Plasma cell leukemia, Waldenstrom macroglobulinemia, POEMS syndrome, or primary AL amyloidosis at the time of screening.
* Subjects who were positive for any of HBsAg, HBV DNA, HCV-Ab, HCV RNA, and HIV-Ab;
* Life-threatening allergic reactions, hypersensitivity reactions, or intolerance to CAR-T cell formulations or their excipients, including DMSO, are known.
* Serious underlying diseases were present.
* Female subjects who were pregnant, breastfeeding, or planning to become pregnant while participating in this study or within 1 year of receiving study treatment.
* Also enrolled in other clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2028-02-20 (Estimated); Study Completion 2029-11-20 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) rate. | From LCAR-F33S cell infusion (Day 1) until the 30th day of follow-up period, assessed up to 30 days
  DLT is classified according to the NCI-CTCAE V5.0 toxicity evaluation criteria and ASTCT consensus classification within 30 days after dose infusion (D1-D30), which is considered by the investigator or collaborator to be reasonably related to LCAR-F33S cell therapy.
Incidence, severity, and type of treatment-emergent adverse events (TEAEs) | From the date of signing ICF to the date 2 years after LCAR-F33S cell infusion
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
To determine the recommended dose for phase II clinical trials (RP2D) | through the last subject of DLT exploration completion, about 2years.
  RP2D was established through accelerated titration design (ATD) and Bayesian Optimal Interval (BOIN) design.
Maximum concentration (Cmax) | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion, assessed about 2 years
  The maximum observed concentration of CAR positive T cells or transgene CAR copy number in peripheral blood.
Time to Cmax | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion, assessed about 2 years
  The time it takes to reach the maximum concentration of CAR positive T cells or transgene CAR copy number in peripheral blood.
Time to the last observed concentration | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion，assessed about 2 years
  The time it takes to reach the last observed concentration of CAR positive T cells or transgene CAR copy number in peripheral blood.
Area Under the Curve (AUC) of the concentration | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion, assessed about 2 years.
  The exposure of CAR positive T cells or transgene CAR copy number in peripheral blood experienced by the subject in a certain time interval.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion, assessed about 2 years
  According to International Myeloma Working Group (IMWG) efficacy criteria. ORR is defined as the proportion of patients with PR or better response after infusion of LCAR-F33S cells.
Very Good Partial Response Rate（VGPR） | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion，assessed about 2 years
  Proportion of subjects achieving VGPR according to IMWG criteria.
Complete response(CR) | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion，assessed about 2 years
  Proportion of subjects achieving CR according to IMWG criteria.
Stringent complete response(sCR) | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion，assessed about 2 years
  Proportion of subjects achieving sCR according to IMWG criteria.
Minimal residual disease (MRD) negative rate | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression, assessed about 2 years
  Proportion of subjects achieving minimal residual disease (MRD) negative rate according to IMWG criteria.
Time-to-response(TTR) | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion, assessed about 2 years
  According to International Myeloma Working Group (IMWG) efficacy criteria. TTR is defined as the interval from the date of the first infusion of the LCAR-F33S cells to the date of the first efficacy assessment for which the subject met all criteria for PR or better. Analyses were performed only in responders.
Duration of response(DOR) | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion，assessed about 2 years.
  According to International Myeloma Working Group (IMWG) efficacy criteria. DOR is defined as the time from the first documented response (PR or better response) to the first documented evidence of disease progression (as defined according to IMWG criteria) or death from any cause.
Progression-free survival(PFS) | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion, assessed about 2 years.
  According to International Myeloma Working Group (IMWG) efficacy criteria. PFS is defined as the interval from the date of the first infusion of the LCAR-F33S cells to the first documentation of disease progression (according to IMWG criteria) or death from any cause, whichever occurred first.
Overall survival(OS) | From the 7th days before first dose of pretreatment with chemotherapy until the date of first documented progression or study completion, assessed about 2 years.
  According to International Myeloma Working Group (IMWG) efficacy criteria. Overall survival (OS) is defined as the interval from the date of the first infusion of LCAR-F33S cells to death.
Occurrence rate of antidrug antibody | From LCAR-F33S cells infusion until the date of first documented progression or study completion, assessed about 2 years.
  Occurrence rate of LCAR-F33S cells preparation ADA.

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, MD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (3):
- China (3):
  - Beijing Boren Hospital, Beijing
  - Institute of Hematology & Blood Diseases Hospital, Tianjin
  - Wuhan Union Hospital, Wuhan

IPD SHARING:
Plan to Share IPD: No